CLINICAL TRIAL: NCT03707340
Title: A Feasibility Study of Flibanserin in Breast Cancer Survivors on Tamoxifen and Aromatase Inhibitors
Brief Title: A Study of Flibanserin in Breast Cancer Survivors on Tamoxifen or Aromatase Inhibitors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-109
Record Dates: First submitted 2018-09-17; First posted 2018-10-16 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Hyposexual Desire Disorder
Keywords: tamoxifen; Flibanserin; hyposexual desire disorder
MeSH Terms: conditions — Breast Neoplasms | interventions — flibanserin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Breast Cancer Pts with hyposexual desire disorder/HSDD (Experimental)
  Interventions: Drug: Flibanserin Pill

INTERVENTIONS:
Drug: Flibanserin Pill — Eligible participants will begin treatment with flibanserin 100 mg orally daily at bedtime for 24-36 weeks and followed for a total of 52 weeks.

SUMMARY:
The purpose of this study is to determine if it is feasible for women to take both Flibanserin and tamoxifen for the duration of the study. This study is also trying to find out if Flibanserin improves or has any effect on hyposexual desire disorder/HSDD in women who are taking tamoxifen for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women age 21 and older
* Able to swallow tablets
* History of stage 0-III breast cancer that is estrogen and/or progesterone receptor positive
* History of breast cancer with no current evidence of disease and have completed primary treatment with any combination of surgery, radiation and/or chemotherapy at least 3 months ago and is currently on Tamoxifen, an AI, or ovarian suppression.
* Has been taking tamoxifen, an AI, ,or ovarian suppression for at least 3 months.
* Has LFTS within 2 times the upper limit of normal proven by a Comprehensive Metabolic Panel (CMP) performed within 6 months of protocol enrollment and while the patient was on Tamoxifen, an AI, or ovarian suppression
* Patients meet criteria for the diagnosis of HSDD as defined by the DSM-IV and ISSWSH Consensus paper. The criteria states that there must be a decrease in sexual desire and this must be a change for at least 3 months from what it was previously. Personal distress resulting from this change must occur. Initial screening will take place with The Decreased Sexual Desire Screener, a 5-question screening tool developed and validated to aid clinicians in making the diagnosis of HSDD. A "yes" response to the first 4 questions on the screener is consistent with HSDD.
* Patients must agree to follow the guidelines for alcohol consumption during the 24 weeks of treatment on study
* English speaking
* Able to participate in the informed consent process

Exclusion Criteria:

* Active secondary cancer requiring cytotoxic chemotherapy
* History or current diagnosis of metastatic breast cancer.
* Unwillingness to follow alcohol guidelines while taking flibanserin
* Hepatic dysfunction (more than 2 times the upper limit of normal for alt, ast, t.bili or alk phos) proven by Comprehensive Metabolic Panel (CMP) performed within 6 months of protocol enrollment and while the patient was on Tamoxifen or an AI
* Patients on strong CYP3A4 inhibitors including ketoconazole, itraconazole, posaconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, boceprevir, telaprevir, telithromycin, conivaptan
* Patients on moderate CYP3A4 inhibitors including Amprenavir, atazanavir, ciprofloxacin, diltiazem, erythromycin, fluconazole, fosamprenavir, verapamil, grapefruit juice
* Non-English speaking
* Unable to participate in the informed consent process

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2026-10-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
Discontinuation rate of flibanserin in women with breast cancer on Tamoxifen with disease or medical induced hypoactive sexual desire disorder | 1 year
  To evaluate the feasibility defined as the treatment discontinuation rate of flibanserin for 24 weeks due to toxicity, withdrawal of consent or other events related to tolerability.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of flibanserin | 1 year
  The AE reporting period begins on the first day of study drug administration and continues until 4 weeks after the patient has taken the last dose of study drug. AE's will be evaluated using CTCAE v 4.

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Norwalk Hospital, Norwalk, Connecticut
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org